CLINICAL TRIAL: NCT06070974
Title: ExosoMe as Integrative Tool for pRognostic Stratification of Adverse Cardiac remodeLing in stEmi Patients: the MIRACLE Study
Acronym: MIRACLE
Status: Recruiting | Type: Observational
Sponsor: Centro Cardiologico Monzino (Other)
Collaborators: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: CCM 1931
Record Dates: First submitted 2023-08-22; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: STEMI
Keywords: Cardiovascular Magnetic Resonance; PCI; Exosome
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood collection for exosome isolation and analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single arm study: STEMI patients, who meet all the inclusion and none of the exclusion criteria, will be enrolled 3 days after PCI to study the correlation between exosome profile and severity of myocardial infarction
  Interventions: Diagnostic Test: CMR and blood collection

INTERVENTIONS:
Diagnostic Test: CMR and blood collection — All patients enrolled will undergo 2 CMR examination (within 3-5 days post PCI and after six months), and blood collection at third day after PCI (T0). Patients recruited at Centro Cardiologico Monzino will be subjected to a blood withdrawal also at different time points: 1- 3- 6 months after STEMI (T1, T2, and T3 respectively).

SUMMARY:
This is a multicenter observational prospective study aimed to assess whether plasma exosomes can help identify, at an early stage, patients at high risk of adverse remodeling after STEMI (ST-elevation myocardial infarction) , thus accelerating proper patient management in order to reduce the risk of future cardiovascular events. In order to study the correlation between exosome profile and severity of myocardial infarction, consecutive STEMI patients will be enrolled 3 days after Percutaneous Coronary Intervention (PCI).

DETAILED DESCRIPTION:
Adverse cardiac remodeling is a process of structural and functional changes associated with worse clinical outcomes and increased mortality, which occurs in response to sustained pathophysiological stimuli, such as ST-elevation myocardial infarction (STEMI). Despite the progresses achieved with reperfusion therapy in STEMI, a significant portion of patients still develops adverse remodeling. Cardiovascular Magnetic Resonance (CMR) is the gold standard for clinical diagnosis of adverse remodeling, as it provides reliable and reproducible information on ventricular size, function and tissue damage. However, CMR is not always applicable, due to resources and availability reasons and to patients' contraindications. Therefore, additional markers for the early detection of patients at risk for adverse remodeling after STEMI are needed. Exosomes are small extracellular vesicles released by cells and detectable in all body fluids, including plasma. Their release and cargo are influenced by cellular microenvironment, thus mirroring cell/organ status. Previous study demonstrated that concentration and cargo of plasma exosomes released during STEMI well reflect the pathophysiology of the disease, suggesting their potential as biomarkers. Whether exosome profile analysis could predict adverse remodeling after STEMI remains to be investigated.

The relevant hypothesis to be tested is whether plasma exosomes may help to identify, in an early phase, patients at high risk of adverse remodeling after STEMI, accelerating proper patient management in order to reduce risk of further cardiovascular events and improve outcomes. Overall, this new knowledge will pave the way toward a new strategy to predict adverse remodeling in STEMI patients and to develop patient-tailored therapy.

ELIGIBILITY:
Inclusion Criteria:

* chest pain suggestive of myocardial ischemia lasting >30 min
* electrocardiogram (ECG) showing ST-segment elevation >0.1 mV in more or equal to 2 limb leads or >0.2 mV in more or equal to 2 contiguous precordial leads, or presumed new left bundle-branch block
* successful treatment with pPCI within 12 h from the onset of symptoms

Exclusion Criteria:

* previous myocardial infarction (MI)
* time to pPCI >12 h
* atrial fibrillation
* renal failure with glomerular filtration <30 ml/min
* claustrophobia
* other contraindications to CMR.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with acute STEMI will be screened for study eligibility by site personnel to identify those who meet all selection criteria
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Verify whether the profile of circulating plasma exosomes reflects CMR-assessed STEMI severity at hospital discharge | within 3-5 days post PCI
  Assess the ability of exosome profile, detected in the blood sample 3 days after PCI (T0),to reflect STEMI severity as assessed by CMR and evaluate the correlation of T0 exosome profile with clinicopathological features.
Evaluate whether exosome profile in the acute phase of hospitalization after STEMI predicts adverse remodeling at six months | 6 months
  Assess the ability of T0 exosomes to predict adverse cardiac remodeling, both alone or in combination with CMR analysis and discover new exosome candidates able to predict adverse cardiac remodeling
Assess whether changes in exosomes profile a different time points following STEMI (1-3-6 months) reflects clinical outcome | 6 months
  Evaluate the change of exosomes profile during time and test the correlation of exosomes change during time or at specific time points with clinical complication and outcome

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Baggiano, MD, Principal Investigator — IRCCS Centro Cardiologico Monzino
Locations (2):
- Italy (2):
  - IRCCS Centro Cardiologico Monzino, Milan, Milan
  - Istituto Auxologico Italiano, Milan

REFERENCES:
- [Background] Pontone G, Carita P, Rabbat MG, Guglielmo M, Baggiano A, Muscogiuri G, Guaricci AI. Role of Cardiac Magnetic Resonance Imaging in Myocardial Infarction. Curr Cardiol Rep. 2017 Aug 31;19(10):101. doi: 10.1007/s11886-017-0907-1. PMID 28856546
- [Background] Masci PG, Pavon AG, Pontone G, Symons R, Lorenzoni V, Francone M, Zalewski J, Barison A, Guglielmo M, Aquaro GD, Galea N, Muscogiuri G, Muller O, Carbone I, Baggiano A, Iglesias JF, Nessler J, Andreini D, Camici PG, Claus P, de Luca L, Agati L, Janssens S, Schwitter J, Bogaert J. Early or deferred cardiovascular magnetic resonance after ST-segment-elevation myocardial infarction for effective risk stratification. Eur Heart J Cardiovasc Imaging. 2020 Jun 1;21(6):632-639. doi: 10.1093/ehjci/jez179. PMID 31326993
- [Background] Kalluri R, LeBleu VS. The biology, function, and biomedical applications of exosomes. Science. 2020 Feb 7;367(6478):eaau6977. doi: 10.1126/science.aau6977. PMID 32029601
- [Background] Zara M, Campodonico J, Cosentino N, Biondi ML, Amadio P, Milanesi G, Assanelli E, Cerri S, Biggiogera M, Sandrini L, Tedesco CC, Veglia F, Trabattoni D, Blandini F, Tremoli E, Marenzi G, Barbieri SS. Plasma Exosome Profile in ST-Elevation Myocardial Infarction Patients with and without Out-of-Hospital Cardiac Arrest. Int J Mol Sci. 2021 Jul 28;22(15):8065. doi: 10.3390/ijms22158065. PMID 34360827